CLINICAL TRIAL: NCT01514084
Title: Cosmetic Outcomes and Patient Satisfaction After Facial Laceration Repair in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1108-081
Record Dates: First submitted 2012-01-12; First posted 2012-01-20 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Facial Lacerations
Keywords: laceration; emergency; cosmetic outcomes; patient satisfaction; suture
MeSH Terms: conditions — Lacerations; Emergencies; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- PEM group: Patients whose lacerations have been repaired by PEM trained physicians.
- GP group: Patients whose lacerations have been repaired by general pediatricians.
- PNP group: Patients whose lacerations have been repaired by PNPs.
- RN group: Patients whose lacerations have been repaired by suture RNs.

SUMMARY:
Facial lacerations are commonly treated in the emergency department. The nature of the injury leads to a great deal of concern about the long-term cosmetic appearance of the wounds.

Research Questions

1. What is the association between wound characteristics, wound management in the ED, patient satisfaction in the ED, and patient-rated cosmetic appearance of sutured wounds?
2. Is there a difference noted among ED providers with different levels of training?
3. Is there an association between initial satisfaction scores and wound outcome?
4. Is there an association between short term and long term wound scores?

Design This is a non-randomized, prospective, observational study of patients who present to the ED seeking treatment for facial laceration repair.

ELIGIBILITY:
Inclusion Criteria:

* Families presenting to the ED for repair of facial laceration will be approached for study inclusion if:

  * Their child seeking treatment is less than 18 years of age
  * The laceration was sustained less than 12 hours prior to presentation to Children's ED
  * They speak English

Exclusion Criteria:

* Families presenting to the ED for repair of facial laceration will be excluded from study participation if they:

  * Are medically complex children
  * Have a history of pre-existing coagulopathy or collagen vascular disease
  * Have a history of immunodeficiency or diabetes mellitus
  * Are suspected of non-accidental trauma
  * Have wounds that could be approximated by tissue adhesives
  * Have animal or human bites
  * Have gross contamination
  * Have puncture wounds
  * Have lacerations of tendon/nerve/cartilage
  * Have scalp lacerations
  * Do not speak English

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric emergency department
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome | 6 months
  Cosmetic Visual Analog Score and the Wound Evaluation Score

SECONDARY OUTCOMES:
Satisfaction score | 6 months
  Visual analog scale; left end labeled "Dissatisified" and right end labeled "Very satisfied"

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Twin Cities, Minnesota, United States

REFERENCES:
- [Background] Quinn JV, Wells GA. An assessment of clinical wound evaluation scales. Acad Emerg Med. 1998 Jun;5(6):583-6. doi: 10.1111/j.1553-2712.1998.tb02465.x. PMID 9660284